CLINICAL TRIAL: NCT00741741
Title: Phase I, Double Blind, Randomized, Placebo-controlled Trial to Examine the Safety, Tolerability and Plasma Pharmacokinetics of Multiple (Monthly) Intramuscular and Subcutaneous Doses of TMC278LA.
Brief Title: TMC278-TiDP15-C150: Trial to Examine Safety, Tolerability and Plasma Pharmacokinetics of Multiple Doses of TMC278LA.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015295
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: HIV-1
Keywords: TMC278-C150; TMC278-TiDP15-C150; HIV-1 infected patients; Intramuscular or subcutaneous injection; Nanosuspension; Therapy; Prevention; Healthy volunteers; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TMC278

SUMMARY:
The purpose of this study is: to determine the safety, (local) tolerability and plasma exposure over time of single intramuscular (IM) doses of 600 and 1200 mg of a new formulation (F006) of TMC278LA, to determine the safety, (local) tolerability and long-term plasma exposure over time of 2 dose regimens of 4 monthly IM doses of a new formulation (F006) of TMC278LA., To determine the safety, (local) tolerability and long-term plasma exposure over time of 1 dose regimen of 4 monthly subcutaneous (SC) doses of a new formulation (F006) of TMC278LA.

DETAILED DESCRIPTION:
Human immunodeficiency virus type 1 (HIV-1)-infected patients are routinely being treated with combinations of 3 or 4 drugs (highly active antiretroviral therapy [HAART]), including nucleoside/nucleotide analogue reverse transcriptase inhibitors (NRTIs/NtRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), and protease inhibitors (PIs), to reduce the risk of viral resistance development. TMC278 is a new potent and selective NNRTI under development. It may be able to prevent replication of the virus and by consequence, prevent new HIV-1 infection. For this novel indication, a sustained release parenteral (IM = Intramuscular or SC = Subcutaneous) formulation, named TMC278LA, allowing sporadic dosing is under development. As a second perspective, the TMC278LA has been designed to cope, for therapeutic treatment in patients, with pill burden and the obligation of having uninterrupted NNRTI treatment at very regular time intervals, imposing considerable compliance constraints on HIV-infected patients. This formulation intends to improve the quality of life of the patient and the drug compliance of the NNRTI treatment. This is a randomized, double-blind (neither patient nor the physician know the name of the study drug), placebo-controlled clinical study to evaluate the safety, (local) tolerability and plasma pharmacokinetics of multiple doses of a novel formulation (nanosuspension) of TMC278LA, containing 300 mg of TMC278 per mL. A total of 30 healthy volunteers will be selected and equally divided into 3 panels. This study will be conducted in male or female volunteers. The clinical study may not necessarily be balanced regarding gender, but it is intended to aim at 50% of each gender. For safety reasons, females must be post-menopausal or surgically sterile. The clinical study consists of 3 panels: Panel 1 (Multiple Dose 1 = MD1), Panel 2 (Multiple Dose 2 = MD2) and Panel 3 (Multiple Dose 3 = MD3). MD1, MD2 and MD3 will receive a multiple dosing regimen of the new formulation of TMC278LA consisting of 4 successive IM doses (at a 1-month interval) in the Gluteus maximus (MD1 and MD2) or 4 successive SC doses (at a 1- month interval) in the periumbilical region (MD3). The first dose (the loading dose) is twice as high as the following 3 doses. Data collected after the first dose in each regimen will serve as a substitute for a single dose. The dosing regimens are: MD1=600/300/300/300 mg; MD2=1200/600/600/600 (IM) and MD3=1200/600/600/600 mg (SC). The study population will include a total of 30 healthy adult volunteers. Ten volunteers will be enrolled in MD1, MD2 and MD3 (6 on active, 2 on vehicle, 2 on saline). Each IM dose will be given at one Injection Site (IS) (in the Gluteus maximus muscle), except for the 1200 mg dose in MD2 for which 600 mg will be injected in each muscle (left and right Gluteus maximus muscle). Likewise, the SC doses will be given at one IS (periumbilical region), except for the 1200 mg loading dose for which 600 mg will be injected in two ISs on either site of the umbilicus. The new formulation has a concentration of 300 mg/mL of TMC278LA. Hence, the maximum volume to be injected per injection site is 2 mL. For the multiple injection panels, rotation of the injected site is recommended. The purpose of the dose sequence in all 3 MD panels is to provide a loading dose for the 300 mg (MD1) and 600 mg (MD2, 3) once monthly regimens. In pharmacokinetics, a loading dose refers to an initial higher dose of a drug that may be given at the beginning of a course of treatment before dropping down to a lower maintenance dose. A first safety review is planned after the first 3 patients and if no acute effects are observed, the following 3 patients will be dosed. A 2nd safety review is planned and if no acute effects are observed, the last 4 patients will be dosed. Within each Panel, the second dose will only be administered when the first dose was considered safe and well tolerated. The first dose of MD2 will start 1 month after start of MD1, when the first IM dose of MD1 has been evaluated in a Data Review Meeting (DRM), approximately 3 weeks after dosing, and is considered safe and well tolerated. Similarly, MD3 will start after the first dose in MD2 is considered safe and well tolerated during a DRM. An extra DRM will be planned approximately 3 weeks after the 4th dose of each panel, in order to evaluate the safety and (local) tolerability after 4 successive doses given at a 1-month interval. Dose Limiting Toxicities and stopping rules will guide decision making during the DRMs. At the DRMs, all safety, local tolerability, systemic tolerability and pharmacokinetic data collected till and including 2 weeks after dosing will be evaluated. Based on these data collected after the loading dose (1st dose), the investigator and the sponsor will decide whether it is safe to proceed to the next dose in a given panel. The next dose can be adjusted, if required, based on safety or pharmacokinetic data available at that time, but will not exceed 600 mg in MD1 and 1200 mg in MD2 and MD3. Such a dose adjustment is applicable to all patients of that particular panel. Upon unblinding on Week 24, patients who were on placebo treatment are allowed to leave the study. In addition, patients who received active treatment and for which the TMC278 plasma concentration in the last sample taken prior to unblinding (= WK20) is below 20 ng/mL are allowed to leave the study as well, provided that there are no persistent AEs that require further follow-up. All patients on active treatment with TMC278 plasma concentrations above 20ng/mL in the last sample taken prior to unblinding, or patients with AEs that require further follow up will be followed up until plasma exposure of TMC278 is below 20 ng/mL or until pending adverse events are resolved or stabilized, respectively. Based on results of the TMC278-TiDP15-C146 clinical study, more than 90% of TMC278 is expected to be washed out within 20 weeks after the last dose. In case TMC278 exposure is still above 20 ng/mL at the WK 32 visit or in case of a persistent AE that needs further follow up, the follow up period will be extended until TMC278 plasma exposure is below 20 ng/mL, or until the AE is resolved or stabilized. The decision to extent the follow-up period will be communicated to the respective subjects at WK33. These patients will be asked to visit the site once every 4 weeks in case of follow-up on TMC278 plasma exposures. Frequency of on-site follow-up on safety will be determined by the investigator on a case by case basis. In this Phase-I study in healthy volunteers no further treatment or medical care is planned after the end of the clinical study. There are 3 panels, and patients will be randomized to treatment with either TMC278LA (n=6), vehicle (n=2) or saline (n=2). The dosing regimens consist of 4 successive doses at a 1-month interval. Dosing regimens are MD1 = 600/300/300/300 mg (IM), MD2 = 1200/600/600/600 mg (IM) and MD3 = 1200/600/600/600 mg (SC). Patients who received saline or vehicle, or who have TMC278 plasma exposures below 20 ng/ml, will leave the study at WK24. Other patients will continue till WK32 or beyond.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 55 years, extremes included
* Non-smokers for at least 3 months prior to selection
* Normal weight as defined by a Body Mass Index (BMI: weight in kg divided by height in meters squared) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form signed voluntarily
* Able to comply with protocol requirements
* Normal 12-lead electrocardiogram (ECG) (in triplicate) at screening including: a) normal sinus rhythm (heart rate [HR] between 40 and 100 bpm), b) QTc interval <= 450 ms, c) QRS interval lower than 120 ms, d) PR interval <= 220 ms
* Healthy on the basis of a pre-study physical examination, medical history, vital signs and the results of blood biochemistry and hematology tests and a urinalysis carried out at screening
* Patient agrees not to participate in any other clinical trial until 6 weeks after being informed that his/her TMC278 exposure is below 20 ng/ml (all panels)
* Females participating in the clinical study must be of non-childbearing potential (e.g. surgically sterilized or postmenopausal with no menstrual bleeding for at least 2 years prior the clinical study
* If the patient is a sexually active man and not surgically sterilized, he must be willing to abstain from sexual intercourse, or use a condom plus another form of contraception (e.g., spermicide, IUD, birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a woman who could become pregnant. This will avoid pregnancy caused by possibly damaged sperm. Males must use a condom during sexual intercourse with pregnant or lactating females. Male patients must not father a child from administration of the first dose and up to one month after the last dose of the IMP.

Exclusion Criteria:

* Past history of heart arrhythmias (extrasystolic, tachycardia at rest) or having baseline prolongation of QTc interval > 450 ms, history of risk factors for Torsade de Pointes syndrome (hypokalemia, family history of long QT Syndrome)
* History or suspicion of alcohol, barbiturate, amphetamine, recreational or narcotic drug use that could impact compliance to protocol requirements and/or safety
* Hepatitis A infection (confirmed by hepatitis A antibody), or hepatitis B infection (confirmed by hepatitis B surface antigen), or hepatitis C infection (confirmed by hepatitis C virus antibody) or HIV-1 or HIV-2 infection at screening
* A positive urine drug test at study screening. Urine will be tested for the presence of amphetamines, benzodiazepines, cocaine, cannabinoids, opioids, methadone and barbiturates
* Currently active or underlying gastro-intestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory or infectious disease
* History of clinically relevant skin disease such as, but not limited to, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria
* History of drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous clinical studies with experimental drugs
* Use of concomitant medication, including over-the-counter products, herbal medication (including St. John's Wort) and dietary supplements, except for paracetamol (acetaminophen) or ibuprofen in a period of 14 days before the first IMP administration
* Participation in an investigational drug trial within 30 days prior to the first injection with IMP, Donation of blood or plasma in the 60 days preceding the injection with the IMP, Having previously participated in a clinical study with oral TMC278 (previously known as R278474) or TMC278LA, Vulnerable subjects (e.g., persons kept in detention)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety, (local) tolerability and TMC278 PK of multiple doses of a novel formulation of TMC278LA throughout the study till WK24, WK28, WK32 or beyond WK32 (i.e. till TMC278 is below 20 ng/ml and till all AEs are resolved/stabilized)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited